CLINICAL TRIAL: NCT07036835
Title: Clinical Investigation of the WaveLight® Ultraviolet Femtosecond Laser for Corneal Flap Creation
Brief Title: Clinical Investigation of a Femtosecond Laser for Corneal Flap Creation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFO268-C009
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Refractive Errors
Keywords: LASIK
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- UV fs-Laser/Anesthetic 1 Right, IR fs-Laser/Anesthetic 1 Left (Other): LASIK surgery performed with the UV fs-Laser (right eye) and IR fs-Laser (left eye) as randomized with Anesthetic 1 eye drops
  Interventions: Procedure: LASIK Surgery; Device: UV fs-Laser; Device: IR fs-Laser; Device: Anesthetic 1 eye drops
- UV fs-Laser/Anesthetic 1 Left, IR fs-Laser/Anesthetic 1 Right (Other): LASIK surgery performed with the UV fs-Laser (left eye) and IR fs-Laser (right eye) as randomized with Anesthetic 1 eye drops
  Interventions: Procedure: LASIK Surgery; Device: UV fs-Laser; Device: IR fs-Laser; Device: Anesthetic 1 eye drops
- UV fs-Laser/Anesthetic 2 Right, IR fs-Laser/Anesthetic 2 Left (Other): LASIK surgery performed with the UV fs-Laser (right eye) and IR fs-Laser (left eye) as randomized with Anesthetic 2 eye drops
  Interventions: Procedure: LASIK Surgery; Device: UV fs-Laser; Device: IR fs-Laser; Device: Anesthetic 2 eye drops
- UV fs-Laser/Anesthetic 2 Left, IR fs-Laser/Anesthetic 2 Right (Other): LASIK surgery performed with the UV fs-Laser (left eye) and IR fs-Laser (right eye) as randomized with Anesthetic 2 eye drops
  Interventions: Procedure: LASIK Surgery; Device: UV fs-Laser; Device: IR fs-Laser; Device: Anesthetic 2 eye drops

INTERVENTIONS:
Procedure: LASIK Surgery — Laser assisted in situ keratomileusis (LASIK) surgery conducted for the purpose of correcting refractive error
Device: UV fs-Laser — WaveLight Ultraviolet Femtosecond Laser used for creating a corneal flap during LASIK surgery
  Other Names: Model 1026
Device: IR fs-Laser — WaveLight FS200 Infrared Femtosecond Laser used for creating a corneal flap during LASIK surgery
  Other Names: Model 1025
Device: Anesthetic 1 eye drops — Topical anesthetic used to numb the surface of the eye
  Arms: UV fs-Laser/Anesthetic 1 Left, IR fs-Laser/Anesthetic 1 Right; UV fs-Laser/Anesthetic 1 Right, IR fs-Laser/Anesthetic 1 Left
Device: Anesthetic 2 eye drops — Topical anesthetic used to numb the surface of the eye
  Arms: UV fs-Laser/Anesthetic 2 Left, IR fs-Laser/Anesthetic 2 Right; UV fs-Laser/Anesthetic 2 Right, IR fs-Laser/Anesthetic 2 Left

SUMMARY:
The purpose of this study is to see how safe the WaveLight Ultraviolet Femtosecond Laser, Model 1026 (UV fs-Laser), is for creating corneal flaps during laser-assisted in situ keratomileusis (LASIK) surgery. This study will be conducted in Australia.

DETAILED DESCRIPTION:
Subjects who qualify to participate will have both eyes treated. Each subject will be randomly assigned to 1 of 2 topical anesthetics (numbing eye drops) and each eye will be randomly assigned to either the UV fs-Laser or the WaveLight FS200 Infrared Femtosecond Laser, Model 1025 (IR fs-Laser).

Subjects will attend a total of 6 scheduled study visits, including a preoperative Screening Visit (Day -45 to -1), a Surgery Visit (Day 0), and 4 postoperative visits at Day 1, Week 1, Month 1, and Month 3/exit, for a total individual duration of participation of approximately 4 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Eligible for LASIK treatment;
* Myopia as specified in the protocol;
* Uncorrected distance visual acuity of greater than or equal to 0.30 logMAR;
* Best corrected distance visual acuity of less than or equal to 0.10 logMAR;
* Presence of clear natural lens (non-cataractous eye);
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* An active implanted device for which laser use may be a contraindication;
* Previous ocular surgery;
* Ocular conditions that may affect subject safety or impact study outcomes;
* Acute or chronic disease or illness that would increase the operative risk or confound the outcomes of the study;
* Current use of medications with known ocular side effects and photosensitivity;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Difference of intended and achieved flap thickness measured at center (i.e., corneal apex) | Month 1
  Optical coherence tomography (OCT), a non-invasive imaging test that uses light waves to take cross-section pictures, will be used to measure the thickness of the cornea. This endpoint is pre-specified for the UV fs-Laser only.
Difference of flap thickness measured between central (i.e., corneal apex) and periphery (i.e., 3 millimeter radius) | Month 1
  Optical coherence tomography (OCT), a non-invasive imaging test that uses light waves to take cross-section pictures, will be used to measure the thickness of the cornea. This endpoint is pre-specified for the UV fs-Laser only.
Ability to lift flap at time of surgery | Day 0 Surgery
  The surgeon will record a response on a questionnaire indicating ability to lift the corneal flap at time of surgery (unable to lift flap / able to lift flap). This endpoint is pre-specified for the UV fs-Laser only.
Ocular adverse events (AEs) related to corneal flap creation with UV fs-Laser and IR fs-Laser | Day 0 Surgery up through Month 3
  An AE is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons. AEs pertaining to corneal flap creation that are attributable to the laser will be recorded.
Flap-related loss of best-corrected distance visual acuity (BCDVA) greater than or equal to 2 lines (greater than or equal to 10 letters logMAR) at 1 month postoperative or later | Month 1 up to Month 3
  Visual acuity will be assessed with correction in place (phoropter or trial frame) at a distance of 4 meters under well-lit conditions using letter charts.
Number of device deficiencies | Day 0 Surgery through Month 3
  A device deficiency is defined as any inadequacy of a medical device with respect to its identity, quality, durability, reliability, usability, safety, or performance.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Surgical, Study Director — Alcon Research, LLC
Locations (1):
- Personaleyes, Sydney, New South Wales, Australia